CLINICAL TRIAL: NCT03082053
Title: A Phase Ib Study of Varlitinib in Japanese Subjects With Advanced or Metastatic Solid Tumours
Brief Title: A Study of Varlitinib in Japanese Subjects With Advanced or Metastatic Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ASLAN Pharmaceuticals (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ASLAN001-010
Record Dates: First submitted 2017-02-02; First posted 2017-03-17 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Advanced or Metastatic Biliary Tract Cancer; Advanced or Metastatic Solid Tumors
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Intervention Model Description: 2 studies of single group in 1 protocol
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study I (Experimental): Varlitinib given as monotherapy to Japanese subjects with advanced or metastatic solid tumors
  Interventions: Drug: varlitinib
- Study II (Experimental): Varlitinib given in combination with capecitabine to Japanese subjects with advanced or metastatic biliary tract cancer
  Interventions: Drug: varlitinib; Drug: capecitabine

INTERVENTIONS:
Drug: varlitinib — IMP
  Other Names: ASLAN001
Drug: capecitabine — Companion Medication
  Other Names: Xeloda
  Arms: Study II

SUMMARY:
The purpose of this study is to explore safety and efficacy of varlitinib administered as monotherapy in Japanese subjects with advanced or metastatic solid tumors, and administered as combination with capecitabine in Japanese subjects with advanced or metastatic biliary tract cancer. Also to evaluate pharmacokinetics (PK) of varlitinib, capecitabine and its metabolite.

ELIGIBILITY:
Inclusion Criteria:

* Study I: Subjects with a solid tumour (excluding haematologic tumors) in advanced or metastatic stage
* Study II: Subjects with advanced (unresectable) or metastatic biliary tract cancer (IHCC, EHCC, gallbladder cancer or ampullary carcinoma)

Exclusion Criteria:

* Subjects with concurrent multiple primary cancers.
* Subjects with a history of (non-infectious) pneumonitis that required steroids or current pneumonitis, or with a history of interstitial lung disease or current interstitial lung disease
* Subjects receiving proton pump inhibitors for established, symptomatic gastro-duodenal ulceration or gastroesophageal reflux disease (including the preventive use)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2017-12-07 (Actual); Study Completion 2018-06-06 (Actual)

PRIMARY OUTCOMES:
The number of patients with a dose limiting toxicity (DLT) in the first treatment cycle | 3 weeks
Determine the DLT(Dose Limiting Toxicity) and MTD(Maximum Tolerated Dose) or Recommended Phase II Dose (RP2D) in Phase I setting. | 52 weeks

SECONDARY OUTCOMES:
Pharmacokinetics: varlinitib, capecitabine and 5-FU metabolites levels in terms of Peak Plasma Concentration (Cmax) | Through, Day 1, Day 3, Day 22
Pharmacokinetics: varlinitib, capecitabine and 5-FU metabolites levels in terms of Area under the plasma concentration-time curve (AUC) from 0 to 12 hours (AUC0-12) | Through, Day 1, Day 3, Day 22
Pharmacokinetics: varlinitib, capecitabine and 5-FU metabolites levels in terms of Minimum (trough) plasma concentration (Cmin) | Through, Day 1, Day 3, Day 22
Pharmacokinetics: varlinitib, capecitabine and 5-FU metabolites levels in terms of Elimination half-life of Phase β (t1/2β) | Through, Day 1, Day 3, Day 22

CONTACTS AND LOCATIONS:
Locations (1):
- ASLAN Selected sites, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No